CLINICAL TRIAL: NCT02175914
Title: Erythromycin as a Novel Therapy Against Familial Adenomatous Polyposis and Sporadic Colorectal Cancer by APC Nonsense Mutation Readthrough.
Brief Title: Erythromycin Treatment for Readthrough of APC Gene Stop Codon Mutations in Familial Adenomatous Polyposis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: michal roll (Other Government)
Responsible Party: Sponsor-Investigator, michal roll, director, R&D Division, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-10-RK-0519-CTIL
Record Dates: First submitted 2012-11-26; First posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: FAP-Familial Adenomatous Polyposis
Keywords: Erythromycin; Familial Adenomatous Polyposis (FAP).; APC gene; nonsense mutations
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Erythromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erythromycin (Experimental): Oral treatment with Erythromycin 500mg twice daily.
  Interventions: Drug: Erythromycin

INTERVENTIONS:
Drug: Erythromycin — Oral Treatment with Erythromycin 500mg, twice daily, for 12 weeks

SUMMARY:
Colorectal cancer (CRC) is a leading cause for cancer related mortality in the western world with a lifetime risk of 6%. Etiology is complex, while genetic background significantly affects the risk. Around one third of all genetic disorders as well as most cases of Familial Adenomatous Polyposis (FAP) and a large proportion of all sporadic CRC cases occur as a result of premature nonsense mutations (creating a stop codon) in an individual's adenomatous polyposis coli (APC) gene. Nonsense mutations are single-point alterations in the DNA that prematurely halt the protein translation process, producing a shortened, nonfunctional protein. In many of these cases, if the cell can be 'persuaded' to ignore the premature stop codon signal, the resulting protein may be able to ameliorate or stop the disease.

Recently, members of the aminoglycoside family of antibiotics have been found to induce ribosomal read-through of nonsense mutations, leading to expression of a full length, functional protein. Investigators have recently shown that members of the aminoglycoside and macrolide antibiotic families can induce read-through of the nonsense mutations in the APC gene and lead to reduced oncogenic phenotypes in CRC cells and in different mice models.

The aim of this project is to determine the ability of the macrolide antibiotic-erythromycin to induce read-through of the nonsense mutations in the APC gene and to induce expression of a full length, functional APC protein in patients suffering from FAP and to tests its effect on adenoma number and size and on desmoid tumors in these patients. The future goal is to maximize the effect of stop-codon suppressors on APC while minimizing side effects.

In this study investigators will select FAP patients which carry APC nonsense mutations, treat them with erythromycin PO for 4-6 months and examine colonic and duodenal adenomas as well as abdominal desmoid tumors, that will be documented before during and after treatment. In parallel, investigators will test polyp, adenoma and desmoid tissue samples as well as blood samples from these patients for changes in expression levels of the APC protein and related oncogenic markers.

Suppression of nonsense mutations within the APC gene should be of benefit for patients suffering from FAP, attenuated FAP or multiple adenomas and for patients with advanced or diffuse CRC. Furthermore, given the rapid progress being made in the identification of different nonsense mutations in human genes that lead to mostly un-curable disease, the identification of clinically approved compounds that suppress nonsense mutations and that can be administered long-term without significant side effects would open new venues in the treatment of genetic human diseases that arise from pre-mature stop codons in important coding sequences.

Immediate goal: establish the ability of erythromycin to read-through APC nonsense mutation in FAP patients. The read-through effect of erythromycin will be clinically tested by counting and measuring the number and size of both colonic and duodenal adenomas before and over treatment and by measuring the size of known desmoid tumors. Samples of the adenomas and desmoid tumors will be tested by western blot, immunofluorescence and immunohistochemistry for restoration of APC expression and changes in oncogenic markers. These experiments should be conducted within 6 month.

Long term objective:

1. Determine the lowest dose of erythromycin that can inhibit growth of colonic neoplasia and CRC in patients expressing a truncated APC protein due to nonsense mutations.
2. Examine the ability of a panel of additional macrolide antibiotics to induce APC nonsense mutation suppression using in-vitro methods. Investigators will focus on macrolide antibiotics that are currently in clinical use and are administrated for long terms. These objectives should take around 6 month and will be conducted in parallel.

ELIGIBILITY:
Inclusion Criteria: only patients from families with APC nonsense stop codon mutation.

* above 18 years old.
* A lack of known sensitivity to ERYTHROMYCIN or other macrolide.
* at the relevant subgroup - existence of polyps in the colon or Ileo-anal pouch that classified as adenomas and the size isn't bigger than 10 mm and there's no high grade dysplasia and that not yet need immediate resection of the colon rectal but just a surveillance.
* In the relevant subgroup- existence of polyps in the duodenum that do not require surgery and aren't bigger than 10 mm and with out high grade dysplasia.
* In the relevant subgroup- a tumor that classified as stomach or pelvic desmoid that not yet need immediate resection and which can be measured by ultrasound or MRI.

Exclusion Criteria:

* below 18 years old.
* sensitivity to ERYTHROMYCIN or other macrolide.
* Ileo-anal pouch without adenomas.
* existence of polyps that are classified as adenomas which are bigger than 10 mm and/or with histological of high grade dysplasia.
* Taking medicines that have interactions with ERYTHROMYCIN such as: Carbamazepine, Cyclosporine, barbiturate, PHENYTOIN, Disopyramide, Lovastatin, Bromocriptine: it is recommended to keep careful attention over their Concentrations in the blood and to match the dose.
* significant personal of familial history of ventricular arrhythmia and/or Long QT interval per ECG, or consumption of drugs that may cause prolonged QT.
* Women who're pregnant and those with lack of judgment won't be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of changes in number and size of adenomas measured by upper endoscopy | After 8,12 weeks and 12 months
  Endoscopic and histological response will be tested by upper and lower endoscopies after 8 ,16-20 weeks and 12 months of treatment.
Evaluation of changes in number and size of adenomas measured by lower endoscopy | After 8,12 weeks and 12 months
  Endoscopic and histological response will be tested by upper and lower endoscopies after 8 ,16-20 weeks and 12 months of treatment.
CT and MRI imaging for desmoids | at the begining of the trail (before treatment) and at the end of the treatment (after 4-6 months).
  Desmoids imaging will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Rina Rosin-Arbeseld, Ph.D., Study Director — Department of Anatomy Sackler Faculty of Medicine, Tel Aviv University.; Revital Kariv, MD., Study Director — Department of Gastroenterol Tel Aviv Medical Center, Sackler Faculty of Medicine, Tel Aviv University.
Locations (1):
- Gastrointestinal malignancies department of gastroentrology & liver disease, Tel Aviv Medical Center, Tel Aviv, Israel